CLINICAL TRIAL: NCT05276557
Title: PyloPlus Urea Breath Test System Pediatric Safety and Efficacy Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ARJ Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ARJ-2022-PED
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Helicobacter Pylori; Safety; Efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Indication for H. pylori testing (Experimental): Walk in basis: Symptomatic patients of H. pylori infection will be enrolled for this study if all acceptance criteria are met. Patients will undergo C13 Urea Breath Test (a single dose of 13C urea at 75mg in powder form, to be dissolved in potable water as the kit indicates) in addition to stool antigen test comparison.
  Interventions: Combination Product: PyloPlus Urea Breath Test System; Diagnostic Test: Stool Antigen Test

INTERVENTIONS:
Combination Product: PyloPlus Urea Breath Test System — System containing a kit containing 13C urea and breath collection bags, and an analyzer to test breath samples pre and post 13C ingestion.
Diagnostic Test: Stool Antigen Test — An antigen test performed via a laboratory to test patients' stool for H. pylori

SUMMARY:
This is a multi-center, non-randomized, open label study. Subjects will be enrolled on a walk-in basis. Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study. All children will be exposed to non-radioactive 13C-Urea with citric acid, and shall submit a stool sample.

Centers will house a PyloPlus UBT Analyzer to document results. PyloPlus Analyzer results shall remain blinded to the investigator and treating physician. No patient management decisions should be made based on the investigational PyloPlus® UBT System.

Treating physician will prescribe a H. Pylori Stool Antigen Test to Stool test at either LabCorp or Quest Diagnostic, for the patient, which will be used for diagnostic purposes by the ordering physician.

Total duration of study is anticipated to be approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 3-17 at the time of visit
* Subject/Legal guardian (and subject when relevant) is willing to sing the Informed Consent/Assent Form
* Naive to H. pylori treatment in the past 4 weeks

Exclusion Criteria:

* Pregnant and/or lactating women
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient of the quality of data
* Participation in other interventional trials
* Allergy to test substrates
* Antibiotics taken within 4 weeks of the testing
* Study subjects shall not consume the following items at least 1 hour prior to the PPUBT test: Mouthwash, Chewing Gum, Carbonated Beverages, Cigarette Smoke, Acetone (to simulate the effect of ketone production that may result from some diets), Alcohol, Food
* Children 12 years and older - to be excluded after a written notification from the sponsor is received at the site that the limit of (approx.) 1/3 of the sample size was achieved for this group

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with recorded adverse events | 24 hours
  Number of participants with recorded adverse events after performing urea breath test

SECONDARY OUTCOMES:
Percentage of Agreement | 7 days
  Percentage of agreement between stool test reference standard and continuous urea breath test in assessing presence or absence of Helicobacter pylori infection

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Dolphin Medical Research, Doral, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Harmony United Research, El Paso, Texas